CLINICAL TRIAL: NCT01674075
Title: Lidocaine Serum Levels in Healthy Adult Volunteers: a Pilot Evaluation of the J-Tip Delivery System
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Padma Gulur, MD, Director of Inpatient Pain Services, Massachusetts General Hospital
Other Study IDs: 2012P001141
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: safety; J-Tip Delivery System; pharmacokinetic profile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adult volunteers: Healthy adult volunteers will be administered a J-Tip to the dorsum of his/her hand.

SUMMARY:
The J-Tip device (National Medical Products, Irvine, CA, USA) is a single-use, needle-free anesthesia delivery system, approximately 10cm long and weighing 9g that allow for the rapid delivery of lidocaine hydrochloride prior to peripheral venous access procedures. First introduced in 2001, it uses compressed carbon dioxide for drug delivery into the subcutaneous space. J-Tip is now approved by the U.S. Food and Drug Administration (FDA) for both children and adults.

Designed for patients with needle anxiety and phobia, several clinical trials (Hollingsworth et al, 2000; Cooper JA et al, 2000) have shown the device to be effective with no significant untoward effects, including in children as young as 3 years old (Zempsky et al, 2008). However, two recent cases of toxic serum lidocaine levels in pediatric patients at Massachusetts General Hospital (MGH) following the use of the J-Tip device is concerning. Both patients were administered local anesthetic using the J-Tip device prior to needle-stick and toxicity screens returned with high levels of lidocaine (>6000 mcg/L).

Currently, there is a limited amount of literature available on the safety profile of the J-Tip Delivery System and no study to date has evaluated serum lidocaine levels following its use, likely on the assumption that systemic absorption from the small amount of lidocaine within the device should be negligible. The two pediatric cases highlighted above, seem to suggest otherwise. The purpose of this pilot study is to assess the safety of the J-Tip device on a small population of healthy adults and to determine if elevated lidocaine levels are present systemically or locally. The primary outcome will be lidocaine serum levels following the administration of the J-Tip device measured at the local site and two distal sites to establish lidocaine serum levels following J-Tip administration. We expect lidocaine levels to be undetectable.

ELIGIBILITY:
Inclusion Criteria-

1. Adults (18-59 years old) without known medical illness
2. Subject has capacity to provide informed consent

Exclusion Criteria-

1. Individuals who have recently received "caine" (dental procedures, topical (orajel) or hydrocortisone/lidocaine cream) will be excluded from the study
2. History of liver or kidney problems
3. Individuals receiving chemotherapeutic agents
4. Individuals with the PORT-A-CATH® Implantable Vascular Access System

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Serum lidocaine concentrations | 1 hour post J-Tip administration
  To evaluate the safety and pharmacokinetics of the J-Tip Delivery system by measuring serum lidocaine concentrations in healthy adult volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Padma Gulur, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States